CLINICAL TRIAL: NCT03474614
Title: Effect of Oral Propranolol on mRNA Expression in Symptomatice Caavernous Malformation
Brief Title: Effect of Oral Propranolol on mRNA Expresssion in Symptomatic Cavernous Malformation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Principal Investigator, Lori Wood, Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-0173-30-12
Record Dates: First submitted 2018-03-05; First posted 2018-03-22 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Cavernous Malformations
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System | interventions — Propranolol; DNA

STUDY DESIGN:
Intervention Model Description: Two groups, intervention and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): A Treatment group of ten (n=10) patients that will receive oral propranolol at a dose of 60mg per day (one 60mg ER capsule per day) for 7- to 10-days prior to surgery plus their usual medications.
  Interventions: Drug: Propranolol; Genetic: DNA and RNA Analysis
- Control Group (Other): A control group of 10 (n=10) patients will receive only their routine medications (no propranolol) during the (-7 to -10 days) preoperative period. A control group (n=10) is required to allow for a semi-quantitative comparison with mRNA and miRNA levels in the treatment group.
  Interventions: Genetic: DNA and RNA Analysis

INTERVENTIONS:
Drug: Propranolol — The medication will be administered so that patient receives a minimum of 7- days and maximum of 10-days of treatment with propranolol prior to planned surgical resection of CCM (routine care)
  Arms: treatment group
Genetic: DNA and RNA Analysis — During the operative procedure, a small sample of the patient's blood will be obtained and small (1 to 2cc) tissue sample from the resected cavernous malformation will be collected. The blood and tissue samples will be labeled and stored for subsequent DNA and RNA analysis

SUMMARY:
This is a single center, randomized, trial that will enroll twenty (n=20) patients with a diagnosis of symptomatic cavernous malformations who are planned candidates for surgical resection by one of the investigators, and who meet all of the inclusion and exclusion criteria. Patients will be randomized into two groups: A Treatment group of ten (n=10) patients that will receive oral propranolol at a dose of 60mg per day (one 60mg ER capsule per day) for 7- to 10-days prior to surgery plus their usual medications, and a Control group of 10 (n=10) patients will receive only their routine medications. Currently, the only active treatment alternative for symptomatic cerebral cavernous malformations is surgery.

A control group is required to allow for a semi-quantitative comparison with mRNA and miRNA levels in the treatment group.

DETAILED DESCRIPTION:
This is a single center, randomized, trial that will enroll twenty (n=20) patients with a diagnosis of symptomatic cavernous malformations who are planned candidates for surgical resection by one of the investigators, and who meet all of the inclusion and exclusion criteria. Patients will be randomized into two groups: A Treatment group of ten (n=10) patients that will receive oral propranolol at a dose of 60mg per day (one 60mg ER capsule per day) for 7- to 10-days prior to surgery plus their usual medications, and a Control group of 10 (n=10) patients will receive only their routine medications. Currently, the only active treatment alternative for symptomatic cerebral cavernous malformations is surgery.

A control group is required to allow for a semi-quantitative comparison with mRNA and miRNA levels in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18-years of age.
2. Clinical and imaging diagnosis of a symptomatic Isolated cavernous malformation or Familial cavernous malformation
3. MRI Imaging Grade Type I or Type II (see Table 1)
4. Patient is considered a candidate for surgical resection of their cavernous malformation
5. Written and informed consent obtained prior to the study enrollment.
6. Negative pregnancy test at time of enrollment for women of child-bearing potential.
7. Heart rate greater than 50 beats per minute
8. Systolic blood pressure > 90 mmHg

Exclusion Criteria:

1. Subject is less than 18-years of age.
2. History of allergy to propranolol or other beta blockers.
3. Patient is already taking another beta blocker for cardiac indications.
4. History of asthma presently requiring any active treatment (oral medications or inhalers).
5. History of cardiac dysfunction (as defined by the New York Heart Association Functional Classification grade II, III or IV).
6. Heart rate < 50 beats per minute
7. Systolic blood pressure < 90 mmHg
8. History of diabetes and currently on any anti-hyperglycemic medication.
9. Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
To measure effects of low-dose oral propranolol on global messenger RNA (mRNA) and microRNA (miRNA) expression in the blood and tissue of patients with CCM | -7 to -10 days until surgery
  compare changes noted in mRNA and miRNA in blood and CCM tissue samples of patients who do and do not receive propranolol preoperatively for CCM

SECONDARY OUTCOMES:
To correlate treatment response to propranolol with the underlying established mutations in cerebral cavernous malformation (CCM) genes. | -7 to -10 days until surgery
  correlate and compare genetic mutations seen in CCM genes in tissue of patients who receive propranolol preoperatively
Record adverse event (tolerance to) related to low-dose oral propranolol (60mg ER once daily) | -7 to -10 days until surgery
  Number of reported adverse events in patients taking propranolol

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zabramski, MD, Principal Investigator — Barrow Brain and Spine
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No